CLINICAL TRIAL: NCT06086262
Title: Hand Grip Strength in Athletic and Non-Athletic Girls at Different Phases of Menstrual Cycle
Status: Completed | Type: Observational
Sponsor: Heba Ahmed Mohamed Ahmed (Other)
Responsible Party: Sponsor-Investigator, Heba Ahmed Mohamed Ahmed, Assisstant Lecturer,MISR University for Science and Technology, Cairo University
Organization: Cairo University (Other)
Other Study IDs: P.T.REC/012/003358
Record Dates: First submitted 2023-09-27; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Grip; Athlete; Non-athlete; Menstrual Cycle
Keywords: Menstrual cycle; Female sex hormones; Athletic female; Power

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Athletic group: twenty basketball and tennis players
  Interventions: Device: Hydraulic hand dynamometer (Jamar, Product model J00105, U.S.A)
- Non athletic group: were recruited from undergraduate students
  Interventions: Device: Hydraulic hand dynamometer (Jamar, Product model J00105, U.S.A)

INTERVENTIONS:
Device: Hydraulic hand dynamometer (Jamar, Product model J00105, U.S.A) — The hydraulic hand dynamometer is a reliable and valid an evaluation tool that's used to measure isometric grip force (hand grip strength) .
  The hydraulic pinch gauge is a reliable and valid an evaluation tool that's used to measure isometric pinch force.
  Other Names: Hydraulic pinch gauge(Jamar, Model 65861, U.S.A)

SUMMARY:
The study was designed as an observational study

DETAILED DESCRIPTION:
The study was designed as an observational case-control study

ELIGIBILITY:
Inclusion Criteria:

- 1. The participant had regular menstrual cycles, which were confirmed by using a calendar for three consecutive menstrual cycles, 2. The participant ages ranged from 16 to 22 years old, 3. The body mass index (BMI) ranged from 18.5 to 25 kg/m2. 4. For athletic group, they had participated in basketball and tennis teams for 3 to 4 years.

5. For non-athletic group, they had a sedentary life without any sport activities.

Exclusion Criteria:

* Participants were excluded from the study if they had:

  1. Irregular menstrual cycle
  2. Pelvic inflammatory diseases, pelvic infection or gynecological diseases.
  3. Any musculoskeletal disorders of Upper extremity or surgery, cardiovascular, pulmonary, neurological or systemic conditions.
  4. Receiving contraceptives or any hormonal therapy.

Ages: 16 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Have regular Menstrual cycle
Study Population: Forty healthy post-pubertal virginal females participated in this study. They were divided into two groups' athletic group of twenty basketball and tennis players and non-athletic group of twenty students. The non-athletic girls were recruited from undergraduate students of Faculty of Physical Therapy, Misr University for science and technology, while the athletic girls were recruited from basketball and tennis teams from Mena Garden City Club, 6 October Club and Shooting Club October.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-11-14 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-04-29 (Actual)

PRIMARY OUTCOMES:
Menstrual cycle phases effect on grips power in athletic girls and non-athletic girls. | From November 2021 to April 2023
  Hydraulic hand dynamometer and Hydraulic pinch gauge devices are used to evaluate the power of hand grips

CONTACTS AND LOCATIONS:
Overall Officials: Aml M Yousef, Professor, Principal Investigator — Cairo University; Hamada M Yousef, Study Director — Cairo University; Elham S Hassan, Teacher, Study Director — Cairo University; Heba A Mohamed, Study Chair — Misr for science and techniology
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided